# ClinicalTrials.gov Protocol Document

Official Title: IC-Growth: Enhancing Post-Traumatic Growth in Cancer Survivors Through

**Group-Based Psychosocial Intervention** 

NCT Number: NCTXXXXXXX

Ethical Committee Approval: March 20th, 2024

Document Date: July 31st, 2025

## **Study Protocol**

# **Study Design**

IC-Growth is a multi-phase, non-pharmacological, randomized controlled trial (RCT) aimed at enhancing post-traumatic growth (PTG) among cancer survivors. The study includes an intervention group and a control group, with participants randomly assigned to either condition. The trial targets three cancer populations: breast, colorectal, and head & neck cancer. The intervention is a structured, manualized group program informed by Acceptance and Commitment Therapy (ACT) principles.

The study is conducted in three phases:

- 1. Preparation Phase: A literature review and expert consultation will inform the development of a novel PTG intervention manual. The manual will be co-developed with academic experts and patient organizations and revised based on feedback.
- 2. Implementation Phase: Participants will be randomly assigned to either the intervention or control group. The intervention will be delivered in small, cancer-specific groups (8–10 participants) over 6–8 weekly sessions lasting 90 minutes each. Control group participants will receive standard oncology follow-up without psychosocial intervention. Due to the nature of the study, it will be open-label (no blinding). Baseline and post-intervention data will be collected.
- 3. Synthesis Phase: Based on study results and stakeholder feedback, recommendations for integrating psychosocial support into oncology care in Greece will be developed. A policy brief will address potential implementation barriers and outline practical solutions.

## **Participants**

Participants will be recruited from two oncology hospitals in Thessaloniki, Greece: Theageneio Cancer Hospital and AHEPA University General Hospital. Eligible participants must:

- Be adults (≥18 years old)
- Have completed scheduled chemotherapy and hospitalization
- Have a diagnosis of breast, colorectal, or head & neck cancer within the past five years

#### Exclusion criteria include:

- Current psychiatric treatment
- Untreated mental health conditions
- Cognitive impairments
- Inability to consent or communicate in Greek
- Cancer recurrence
- Diagnosis of a different cancer in the past 5 years
- Life expectancy <12 months

Randomization will be performed via specialized software developed by the Centre for Research and Technology Hellas (CERTH), ensuring strict allocation concealment.

#### Intervention

The intervention will focus on promoting PTG using structured sessions grounded in ACT. Topics include psychological flexibility, mindfulness, narrative reconstruction, meaning-making, and value-based goal setting. Sessions will be led by a trained facilitator and a cofacilitator as needed. Participant feedback will be gathered post-intervention.

## **Statistical Analysis Plan**

#### **Software**

All analyses will be conducted using SPSS version 23.

## **Preliminary Data Handling**

- Outliers and data normality will be examined.
- Reliability of all instruments will be assessed using Cronbach's alpha.
- Demographic and clinical data will be reported using descriptive statistics.

## **Primary Analysis**

The primary outcome—Post-Traumatic Growth (PTG)—will be analyzed using:

- Paired t-tests within groups (pre- vs. post-intervention)
- Independent t-tests or ANCOVA to compare intervention and control groups, adjusting for baseline PTG scores.

### **Secondary Outcomes**

Secondary outcomes will be analyzed similarly:

- Quality of Life and Spiritual Well-being (FACIT-Sp, FACT subscales)
- Anxiety and Depression (HADS)
- Trauma-Related Distress (IES-R)
- Illness Perceptions (BIPQ)
- Salivary Cortisol (biomarker analysis)

Group comparisons will use independent t-tests or ANOVA for continuous variables, chisquare tests for categorical variables, and non-parametric tests as appropriate.

## **Multivariate and Predictive Analysis**

- Multiple regression analyses will explore baseline predictors of PTG and intervention response.
- Factor analysis will examine the structure of PTG domains within the Greek population.
- Exploratory network analysis may identify interactions among psychological and biological variables.

## Sample Size Estimation

Power calculations (via G\*Power 3) determined a minimum of 70–80 participants per group, totaling 140–160 participants, to detect moderate effect sizes with adequate power

( $\beta$  = 0.80) and  $\alpha$  = 0.05. Power analysis was informed by Robson & McCartan (2016) to reduce the risk of Type I and II errors.